CLINICAL TRIAL: NCT05254457
Title: A Multi-Center, Open-Label, Extension Study to Evaluate the Long-Term Safety, Efficacy, and Durability of EN3835 in the Treatment and Retreatment of Plantar Fibromatosis
Brief Title: Long-Term Safety, Efficacy, and Durability of EN3835 in the Treatment and Retreatment of Plantar Fibromatosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-306
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Plantar Fibromatosis
MeSH Terms: conditions — Fibromatosis, Plantar

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Observation Only Group (No Intervention)
- Treated or Retreated Group (Experimental)
  Interventions: Biological: EN3835

INTERVENTIONS:
Biological: EN3835 — Treatment or retreatment with EN3835
  Arms: Treated or Retreated Group

SUMMARY:
Assess the long-term safety and efficacy of EN3835 in participants who have participated in a parent placebo-controlled study of EN3835 (EN3835-222, NCT05152173) and assess the efficacy and safety of EN3835 in the treatment and retreatment of plantar fibromatosis.

ELIGIBILITY:
Inclusion Criteria:

1. Have been enrolled and completed a sponsored-clinical study of EN3835 (for the EN3835-222 study, participants who completed the study are those that completed the Day 57 visit, were assessed for safety and received at least 1 dose of study intervention).
2. Willing and able to comply with all protocol required visits and assessments.
3. Agree not to use opioids during the study period and has not used opioids 2 weeks prior to the Observational Day 1 Visit.
4. Agree to not initiate or change use of orthotics or inserts designed to relieve symptoms of plantar fibromatosis during the study period.
5. Willing and able to comply with all protocol required visits and assessments.
6. Be adequately informed and understand the nature and risks of the study and be able to provide consent
7. If female, be of non-childbearing potential (history of hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or postmenopausal with no history of menstrual flow in the 12 months prior to the Day 1 Visit), or, if of childbearing potential, be nonpregnant, non-lactating and agree to use effective contraception when with a male partner for the duration of the study and for 28 days after any active treatment period.
8. Have no significant medical history or examination findings related to the participant's plantar nodules, which in the investigator's opinion, would make the participant unsuitable for EN3835 administration.

Exclusion Criteria:

1. Has any musculoskeletal, neuromuscular, neurosensory, or other neurological or related disorder that affects the participant's use of his or her feet and/or would impair his/her completion of study assessments as determined by the investigator.
2. Any other significant medical condition or had an SAE in the parent study which in the investigator's opinion, would make the participant unsuitable for enrollment in the study.
3. Received or plans to receive surgical or non-surgical treatments on the foot or nodules that were treated.
4. Has a known systemic allergy to collagenase or any other excipient of EN3835.
5. Has a known bleeding disorder that would make the participant unsuitable for treatment or retreatment in the study.
6. Has significant medical history or examination findings related to the participant's plantar nodules, which in the investigator's opinion, would make the participant unsuitable for EN3835 administration.
7. Has a known coagulation disorder or is taking any medications that would increase the risk of bleeding (except <150mg of aspirin daily, 7 days prior to first injection and for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants reporting adverse events (AE) | Day 1 to Day 450
  Proportion of participants reporting AE during the study assessed by incidence, severity and duration

SECONDARY OUTCOMES:
Change from baseline on the Foot Function Index (FFI) total score in participants treated in the parent studies, and participants retreated in this study | Observational Days 60, 120, 180, 270, 360, and 450
  Change from baseline on the FFI total score on a 5-point rating scale (0-4). This score is comprised of activity limitation, difficulty, and pain subscales. Each subscale is scored on a 5-point rating scale, ranging from 0 to 4, with 0 being never, no difficulty, or none and 4 being always, a lot of difficulty, and extreme.
Change from baseline on the Foot Function Index (FFI) subscales in participants treated in the parent studies, and participants retreated in this study | Observational Days 60, 120, 180, 270, 360, and 450
  Change from baseline on the FFI subscales (pain, difficulty, and activity limitation). This score is comprised of activity limitation, difficulty, and pain subscales. Each subscale is scored on a 5-point rating scale, ranging from 0 to 4, with 0 being never, no difficulty, or none and 4 being always, a lot of difficulty, and extreme.
Change from baseline in the nodular hardness in participants treated in the parent studies, and participants retreated in this study | Observational Days 60, 120, 180, 270, 360, and 450
  Change from baseline in the nodular hardness of the treated nodules measured by durometer
Change from baseline in the nodular consistency of the treated nodules by palpation in participants treated in the parent studies, and participants retreated in this study | Observational Days 60, 120, 180, 270, 360, and 450
  Change from baseline in the nodular consistency of the treated nodules by palpation
Change from baseline on the Pain Intensity Numerical Rating Scale (NRS) in the parent studies, and participants retreated in this study | Observational Days 60, 120, 180, 270, 360, and 450
  Change from baseline on the Pain Intensity NRS ranging from 0 (No Pain) to 10 (Worst Pain Imaginable)
Proportion of participants that meet Treatment Session 1 criteria in the parent studies, and participants retreated in this study | Days 180 or 270
  Proportion of participants that meet Treatment Session 1 criteria
Proportion of participants on the Subject Satisfaction with Treatment Scale in the parent studies, and participants retreated in this study | Observational Days 60, 120, 180, 270, 360, and 450
  Proportion of participants reporting "Quiet Satisfied" (+1) and "Very Satisfied" (+2) on the Subject Satisfaction with Treatment Scale
Proportion of participants on the Clinician Global Impression of Change Scale in the parent studies, and participants retreated in this study | Observational Days 60, 120, 180, 270, 360, and 450
  Proportion of participants reporting "Minimally Improved" (+1), "Much Improved" (+2) or "Very Much Improved" (+3) on the Clinician Global Impression of Change Scale
Change from baseline (Retreatment) on the Foot Function Index (FFI) total score in the parent studies, and participants retreated in this study | Change from baseline (Retreatment Day 1) to Retreatment Days 15, 29,43, 57, 117, 197, and 237
  Change from baseline (Retreatment Day 1) with EN3835 on the FFI total score on a 5-point rating scale (0-4). This score is comprised of activity limitation, difficulty, and pain subscales. Each subscale is scored on a 5-point rating scale, ranging from 0 to 4, with 0 being never, no difficulty, or none and 4 being always, a lot of difficulty, and extreme.
Change from baseline (Retreatment) on the Foot Function Index (FFI) subscales (pain, difficulty, and activity limitation) in the parent studies, and participants retreated in this study | Change from baseline (Retreatment Day 1) to Retreatment Days 15, 29,43, 57, 117, 197, and 237
  Change from baseline (Retreatment Day 1) with EN3835 on the FFI subscales (pain, difficulty, and activity limitation). This score is comprised of activity limitation, difficulty, and pain subscales. Each subscale is scored on a 5-point rating scale, ranging from 0 to 4, with 0 being never, no difficulty, or none and 4 being always, a lot of difficulty, and extreme.
Change from baseline (Retreatment) in the nodular hardness of the treated nodules in the parent studies, and participants retreated in this study | Change from baseline (Retreatment Day 1) to Retreatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Retreatment Day 1) with EN3835 in the nodular hardness of the treated nodules measured by durometer
Change from baseline (Retreatment Day 1) in the nodular consistency of the treated nodules by palpation in the parent studies, and participants retreated in this study | Change from baseline (Retreatment Day 1) to Retreatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Retreatment Day 1) with EN3835 in the nodular consistency of the treated nodules by palpation
Change from baseline (Retreatment Day 1) on the Pain Intensity Numerical Rating Scale (NRS) in the parent studies, and participants retreated in this study | Change from baseline (Retreatment Day 1) to Retreatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Retreatment Day 1) with EN3835 on the Pain Intensity NRS ranging from 0 (No Pain) to 10 (Worst Pain Imaginable)
Proportion of participants reporting on the Subject Satisfaction with Treatment Scale in the parent studies, and participants retreated in this study | Retreatment Days 15, 29, 43, 57, 117, 197, and 237
  Proportion of participants reporting to be "Quiet Satisfied" (+1) and "Very Satisfied" (+2) on the Subject Satisfaction with Treatment Scale on Retreatment Days
Proportion of participants reporting on the Clinician Global Impression of Change Scale in the parent studies, and participants retreated in this study | Retreatment Days 15, 29, 43, 57, 117, 197, and 237
  Proportion of participants reporting "Minimally Improved" (+1), "Much Improved (+2)" or "Very Much Improved (+3) on the Clinician Global Impression of Change Scale on Retreatment Days
Change from baseline (Treatment Day 1) on the Foot Function Index (FFI) total score in the parent studies, and participants retreated in this study | Change from baseline (Treatment 1) to Treatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Treatment Day 1) with EN3835 on the FFI total score on a 5-point rating scale (0-4). This score is comprised of activity limitation, difficulty, and pain subscales. Each subscale is scored on a 5-point rating scale, ranging from 0 to 4, with 0 being never, no difficulty, or none and 4 being always, a lot of difficulty, and extreme.
Change from baseline (Treatment Day 1) on the Foot Function Index (FFI) subscales in the parent studies, and participants retreated in this study | Change from Baseline (Treatment 1) to Treatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Treatment Day 1) with EN3835 on the FFI subscales (pain, difficulty, and activity limitation). This score is comprised of activity limitation, difficulty, and pain subscales. Each subscale is scored on a 5-point rating scale, ranging from 0 to 4, with 0 being never, no difficulty, or none and 4 being always, a lot of difficulty, and extreme.
Change from baseline (Treatment Day 1) in the nodular hardness of the treated nodules in the parent studies, and participants retreated in this study | Change from baseline (Treatment Day 1) to Treatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Treatment Day 1) with EN3835 in the nodular hardness of the treated nodules measured by durometer
Change from baseline (Treatment Day 1) in the nodular consistency of the treated nodules in the parent studies, and participants retreated in this study | Change from baseline (Treatment Day 1) to Treatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Treatment Day 1) with EN3835 in the nodular consistency of the treated nodules be palpation
Change from baseline (Treatment Day 1) on the Pain Intensity Numerical Rating Scale (NRS) in the parent studies, and participants retreated in this study | Change from baseline (Treatment Day 1) to Treatment Days 15, 29, 43, 57, 117, 197, and 237
  Change from baseline (Treatment Day 1) with EN3835 on the Pain Intensity NRS ranging from 0 (No Pain) to 10 (Worst Pain Imaginable)
Proportion of participants reporting on the Subject Satisfaction with Treatment Scale in the parent studies, and participants retreated in this study | Treatment Days 15, 29, 43, 57, 117, 197, and 237
  Proportion of participants reporting to be "Quite Satisfied" (+1) and "Very Satisfied" (+2) on the Subject Satisfaction with Treatment Scale
Proportion of participants reporting on the Clinician Global Impression of Change Scale in the parent studies, and participants retreated in this study | Treatment Days 15, 29, 43, 57, 117, 197, and 237
  Proportion of participants reporting "Minimally Improved" (+1 ), "Much Improved" (+2) or "Very Much Improved" (+3) on the Clinician Global Impression of Change Scale
Presence of anti-AUX-I and anti-AUX-II antibody titer levels | Retreatment/Treatment Day 57 and Day 450
  Presence of anti-AUX-I and anti-AUX-II antibody titer levels in EN3835 treated and retreated participants
Presence of neutralizing antibodies to AUX-I and AUX-II | Retreatment/ Treatment Day 57 and Day 450
  Presence of neutralizing antibodies to AUX-I and AUX-II in EN3835 treated and retreated participants

CONTACTS AND LOCATIONS:
Overall Officials: Nina Green, Study Director — Endo Pharmaceuticals
Locations (27):
- United States (27):
  - Endo Clinical Trial Site #12, Bakersfield, California
  - Endo Clinical Trial Site #3, Fresno, California
  - Endo Clinical Trial Site #23, La Mesa, California
  - Endo Clinical Trial Site #13, Tarzana, California
  - Endo Clinical Trial Site #15, Vista, California
  - Endo Clinical Trial Site #18, Whittier, California
  - Endo Clinical Trial Site #24, Miami, Florida
  - Endo Clinical Trial Site #8, Pinellas Park, Florida
  - Endo Clinical Trial Site #21, Sweetwater, Florida
  - Endo Clinical Trial Site #22, Lawrenceville, Georgia
  - Endo Clinical Trial Site #25, Meridian, Idaho
  - Endo Clinical Trial Site #19, Decatur, Illinois
  - Endo Clinical Trial Site #2, O'Fallon, Illinois
  - Endo Clinical Trial Site #14, Springfield, Illinois
  - Endo Clinical Trial Site #6, Pasadena, Maryland
  - Endo Clinical Trial Site #16, Jefferson City, Missouri
  - Endo Clinical Trial Site #9, York, Pennsylvania
  - Endo Clinical Trial Site #4, Bedford, Texas
  - Endo Clinical Trial Site #17, Dallas, Texas
  - Endo Clinical Trial Site #26, Dallas, Texas
  - Endo Clinical Trial Site #5, Fort Worth, Texas
  - Endo Clinical Trial Site #27, Georgetown, Texas
  - Endo Clinical Trial Site #7, Houston, Texas
  - Endo Clinical Trial Site #10, Houston, Texas
  - Endo Clinical Trial Site #1, McAllen, Texas
  - Endo Clinical Trial Site #11, Salt Lake City, Utah
  - Endo Clinical Trial Site #20, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP